CLINICAL TRIAL: NCT06150170
Title: Evaluation of the Efficiency of Propioceptive Study According to Radiological Stages in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Sibel Gayretli Atan, Physiotherapist, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBU
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; rehabilitation; exercise; physiotherapy; propioception
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): This group includes patients with grade 1 and grade 2 knee osteoarthritis.
  Interventions: Other: Proprioceptive training
- Group 2 (Experimental): This group includes patients with grade 3 and grade 4 osteoarthritis.
  Interventions: Other: Proprioceptive training

INTERVENTIONS:
Other: Proprioceptive training — Proprioceptive exercises were applied to both groups. In addition to these exercises, balance, coordination and strengthening exercises will also be applied to both groups.

SUMMARY:
Evaluation of the Efficiency of Propioceptive Study According to Radiological Stages in Patients with Knee Osteoarthritis

DETAILED DESCRIPTION:
Investigators divided patients with knee osteoarthritis into two groups. Group 1 consisted of stage 1 and stage 2 patients. Group 2 consisted of stage 3 and stage 4 patients. Proprioceptive training was applied in both groups. Investigators aim is to evaluate the effect of proprioceptive exercises on knee osteoarthritis according to the radiological level.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee osteoarthritis by a specialist physician using MRI, US or radiography and physical examination.
* Being between the ages of 35-70
* Stage 1-2-3-4 according to Kellegran Lawrence (K-L) in radiological examination

Exclusion Criteria:

Having active synovitis

* Having received physical therapy in the last 6 months
* Those with neurological problems that affect walking
* Those with serious respiratory, central, peripheral, vascular and uncontrolled metabolic problems that will prevent exercise
* Has had lower extremity surgery in the past
* Intra-articular steroid injections within the last 6 months
* Using psychoactive drugs
* Those with serious vision, hearing and speech disorders
* Patients with vestibular dysfunction will not be included in the study

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Evaluation will be performed before treatment and after 4 weeks rehabilitation program.
  The scale consists of 3 main headings and 24 questions. It is scored between 0 and 100. There is a negative correlation between scoring and functionality.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | Evaluation will be performed at Baseline (before treatment) and 4 weeks
  The levels of pain is felted at rest / activity / night will be measured using Visual Analogue Scale (VAS)..Patients will be asked to evaluate their pain status with a 10-point scale and high scores are positively correlated with pain
Pressure Pain Threshold Measurement | Evaluation will be performed at Baseline (before treatment) and 4 weeks
  A digital algometer will be used for Pressure Pain Threshold Measurement. Digital algometer is a device that objectively evaluates the pressure pain threshold. Low values indicate increased sensitivity and pain sensation.
Range of Motion (ROM) | Evaluation will be performed at Baseline (before treatment) and 4 weeks
  Knee,food and hip ROM will be evaluated with digital goniometer while the patient will be in supine and prone position.
Timed Up and Go Test (TUG) | Evaluation will be performed at Baseline (before treatment) and 4 weeks
  The scale consists of 7 questions measuring the physical activity of the individual in the last 7 days. The activity level is determined according to the scale score.
Manual Muscle Test | Evaluation will be performed at Baseline (before treatment) and 4 weeks
  Manual Muscle Test is a procedure for the evaluation of strength of individual muscle or muscles group, based upon the effective performance of a movement in relation to the forces of gravity or manual resistance through the available ROM.
Short Form 36 (SF-36) | Evaluation will be performed at Baseline (before treatment) and 4 weeks
  SF-36 will be used to assess physical and mental health-related quality of life. The total score is at least 0 and at most 100, and the high scores are positively correlated with high quality of life.
Global Rating of Change (GRC) Scale | 4 weeks
  Global Rating of Change (GRC) scale will be used to assess the overall satisfaction levels of the patients. Patients will be asked to evaluate their post-treatment status with a 5-point likert scale and high scores are positively correlated with satisfaction.
International Physical Activity Scale (IPAQ) | Evaluation will be performed at Baseline (before treatment) and 4 weeks
  The scale consists of 7 questions measuring the physical activity of the individual in the last 7 days. The activity level is determined according to the scale score.
Proprioception Sense | Evaluation will be performed at Baseline (before treatment) and 4 weeks
  The sense of proprioception will be measured using a digital goniometer. It will be repeated 3 times. The average will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Sibel Gayretli Atan, Principal Investigator — sssibel_38@hotmail.com
Locations (1):
- Istanbul Health Sciences University, Üsküdar, Istanbul, Turkey (Türkiye)